CLINICAL TRIAL: NCT04683575
Title: Distribution of Selenium in Patients With Differentiated Thyroid Carcinoma and Effect of Selenium Supplement on Prognosis of Patients With Differentiated Thyroid Carcinoma.
Brief Title: Clinical Study on the Effect of Selenium Yeast Capsule on Prognosis of Differentiated Thyroid Carcinoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Lili Cao, Professor, Qianfoshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XYJA2020
Record Dates: First submitted 2020-11-26; First posted 2020-12-24 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Selenium Deficiency; Thyroid Cancer TNM Staging; Recurrence; Metastasis
Keywords: Selenium; Thyroid Cancer; recurrence; metastasis
MeSH Terms: conditions — Recurrence; Neoplasm Metastasis; Thyroid Neoplasms

STUDY DESIGN:
Intervention Model Description: experimental group：Selenium yeast treatment group control group：Placebo control group blank control group
Who Masked: Participant, Investigator
Masking Description: All participants, investigators were blinded to the grouping of the experiment and the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- experimental group (Experimental): Patients with differentiated thyroid carcinoma with low blood selenium are treated with selenium yeast（dosage form：capsule dosage：200μg bid duration: 5 years）.
  Interventions: Drug: Selenium Yeast
- Placebo control group (Placebo Comparator): Patients with differentiated thyroid cancer with low blood selenium are given placebo treatment（dosage form：capsule dosage：200μg bid duration: 5 years）
  Interventions: Drug: Placebo
- No intervention group (No Intervention): Patients with differentiated thyroid cancer with low blood selenium are not treated.

INTERVENTIONS:
Drug: Selenium Yeast — oral medication
  Arms: experimental group
Drug: Placebo — oral medication
  Arms: Placebo control group

SUMMARY:
Oxidative stress is involved in the pathogenesis of thyroid cancer, but the mechanism is not clear. The thyroid is the organ with the most abundant selenium content, and selenium may be involved in protecting the gland from the influence of large amounts of H2O2 produced during thyroid hormone biosynthesis.

Selenium may exert anti-tumor activity through a variety of mechanisms, including inducing apoptosis and anti-oxidation to change the DNA methylation state of tumor suppressor genes, cell cycle arrest and stimulation of the immune system, as well as playing an anti-tumor role through its anti-inflammatory and anti-angiogenesis properties.

The whole blood and thyroid selenium concentrations in patients with thyroid cancer were lower, and the decreased serum selenium levels were also associated with the high TNM stage of thyroid cancer.

According to the Nutrition Prevention of Cancer (NPC) trial, selenium yeast supplements with a daily selenium content of 200 MCG have been shown to reduce the incidence of total cancer, prostate cancer, colon cancer, and lung cancer, and cancer mortality. The active agent in selenium yeast supplements is known as selenium methionine (SEMET).

In general, the association between selenium and thyroid cancer is still inconclusive, the question of whether low selenium is a predisposition factor or a consequence of thyroid cancer has not been resolved, and the clinical effect of selenium supplementation in preventing thyroid cancer or improving its prognosis remains to be studied.

The hypothesis is that supplementation with selenium yeast will improve the prognosis of patients with differentiated alpha-carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Participants have signed informed consent forms；
2. Patients with differentiated thyroid carcinoma diagnosed pathologically after thyroid surgery；
3. Male or female patients aged 18-75 years;
4. Women who are likely to become pregnant must use the appropriate contraceptive method to avoid pregnancy and minimize the likelihood of conception between the beginning of the drug intervention study and the 28th day after the study.

Exclusion Criteria:

1. A patient who is pregnant or breastfeeding;
2. Currently, hepatase cytochrome P450 3A4 induction or inhibitor therapy, antiviral therapy for immunodeficiency diseases (note: hepatase induction or inhibitor: phenobarbital phenobarbital sodium rifampicin carbamazepine grisoflomycin and dexamethasone and chloramphenicol allopurinol ketone conazole isoniazid imittidine phenothiazine);
3. Gastrointestinal surgery that may affect the study of drug absorption;
4. The patient has a history of haemoglobin disease or acute progressive nephropathy or autoimmune skin disease;
5. A history of substance abuse and alcohol abuse within the last 1 year;
6. There are therapeutic contraindications with selenium yeast capsules as listed in the instructions;
7. New York Heart Association (NYHA) class III or IV congestive heart failure and/or left ventricular ejection fraction of 40% with a significant cardiovascular history in the past 6 months: myocardial infarction coronary angioplasty or bypass surgery valvular disease or repair of unstable angina transient ischemic attack or cerebrovascular accident;
8. There are obvious abnormalities in liver function;
9. The patient has significant liver disease acute active hepatitis or chronic active hepatitis clinical signs or symptoms；
10. Laboratory and physical examination or ECG findings of any clinically significant abnormality would, in the investigator's judgment, compromise the patient's safety or prevent successful participation in the clinical study；
11. Patients with severe renal insufficiency.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2022-05-30 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
recurrence rate | 5 years
  Percentage

SECONDARY OUTCOMES:
metastasis Rate | 5 years
  Percentage

CONTACTS AND LOCATIONS:
Overall Officials: Lin Liao, Doctor, Principal Investigator — Qianfoshan Hospital, The First Hospital affiliated of Shandong First Medical University
Locations (1):
- The First affiliated hospital of Shandong First Medical University, Jinan, Shandong, China

REFERENCES:
- [Background] Gheorghiu ML, Badiu C. Selenium involvement in mitochondrial function in thyroid disorders. Hormones (Athens). 2020 Mar;19(1):25-30. doi: 10.1007/s42000-020-00173-2. Epub 2020 Jan 20. PMID 31960358
- [Background] Metere A, Frezzotti F, Graves CE, Vergine M, De Luca A, Pietraforte D, Giacomelli L. A possible role for selenoprotein glutathione peroxidase (GPx1) and thioredoxin reductases (TrxR1) in thyroid cancer: our experience in thyroid surgery. Cancer Cell Int. 2018 Jan 15;18:7. doi: 10.1186/s12935-018-0504-4. eCollection 2018. PMID 29371830
- [Background] Jonklaas J, Danielsen M, Wang H. A pilot study of serum selenium, vitamin D, and thyrotropin concentrations in patients with thyroid cancer. Thyroid. 2013 Sep;23(9):1079-86. doi: 10.1089/thy.2012.0548. Epub 2013 Jul 17. PMID 23350941
- [Background] Moncayo R, Kroiss A, Oberwinkler M, Karakolcu F, Starzinger M, Kapelari K, Talasz H, Moncayo H. The role of selenium, vitamin C, and zinc in benign thyroid diseases and of selenium in malignant thyroid diseases: Low selenium levels are found in subacute and silent thyroiditis and in papillary and follicular carcinoma. BMC Endocr Disord. 2008 Jan 25;8:2. doi: 10.1186/1472-6823-8-2. PMID 18221503
- [Background] Marshall JR, Burk RF, Payne Ondracek R, Hill KE, Perloff M, Davis W, Pili R, George S, Bergan R. Selenomethionine and methyl selenocysteine: multiple-dose pharmacokinetics in selenium-replete men. Oncotarget. 2017 Apr 18;8(16):26312-26322. doi: 10.18632/oncotarget.15460. PMID 28412747
- [Background] Barrea L, Gallo M, Ruggeri RM, Giacinto PD, Sesti F, Prinzi N, Adinolfi V, Barucca V, Renzelli V, Muscogiuri G, Colao A, Baldelli R; E.O.L.O. Group. Nutritional status and follicular-derived thyroid cancer: An update. Crit Rev Food Sci Nutr. 2021;61(1):25-59. doi: 10.1080/10408398.2020.1714542. Epub 2020 Jan 30. PMID 31997660